CLINICAL TRIAL: NCT03180853
Title: Multiple Myeloma Patient Registry
Status: Terminated | Type: Observational
Why Stopped: Completion of study in orig timeframe not feasible considering evolving treatments for MM in US.
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108326; NOPRODMMY4001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsed Multiple Myeloma Participants: The participants in the United States with a confirmed diagnosis of relapsed multiple myeloma following 1 to 3 prior lines of therapy who initiate treatment with a proteasome inhibitor (PI) and/or immunomodulatory drug (IMiD) used either as monotherapy or combination therapy with other treatments as per routine clinical practice within 90 days prior to study enrollment. These participants will be observed for the sequence of systemic myeloma treatments used during routine clinical practice, considering the life expectancy of patients with myeloma in the registry.

SUMMARY:
The purpose of this study is to document the participants characteristics, disease burden, and clinical management of participants in the United States who are treated for relapsed multiple myeloma in routine medical practice with a treatment strategies that include a proteasome inhibitor (PI) and/or immunomodulatory drug (IMiD) used either as monotherapy or combination therapy with other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must sign, and/or their legally acceptable representative where applicable must sign, a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements
* Have a diagnosis of relapsed MM [according to 2014 International Myeloma Working Group (IMWG) criteria] with 1 to 3 prior lines of therapy. (An induction regimen followed by autologous stem cell transplantation and single-agent maintenance therapy will be considered a single line of therapy.)
* Participants must have initiated a new line of induction therapy that includes a proteasome inhibitor (PI) and/or immunomodulatory drug (IMiD) within 90 days prior to enrollment. A short course of corticosteroids is allowed prior to initiating the new line of induction therapy
* Must be willing and able to complete the protocol-required patient-reported outcome (PROs)

Exclusion Criteria:

* Participant has plasma cell leukemia [greater than (>) 2.0 * 10^9 per liter] circulating plasma cells by standard differential), Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and/or skin changes), or amyloid light-chain amyloidosis
* Participant has a life expectancy of less than 6 months
* At the time of screening, participant is enrolled in an interventional clinical trial for MM using an anti-neoplastic agent that is not currently approved by the United States (US) Food and Drug Administration (FDA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants to be enrolled in this registry will be participants whose multiple myeloma (MM) has relapsed after the administration of 1 to 3 prior lines of therapy and who initiate treatment with a proteasome inhibitor (PI) and/or immunomodulatory drug (IMiD) used either as monotherapy or combination therapy with other treatments within 90 days prior to study enrollment. Participants are to be recruited from medical centers in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 3 years
  Overall response rate defined as the percentage of participants achieving Complete Response (CR), Very good partial response (VGPR), or Partial response (PR) (CR + VGPR + PR) as per International Myeloma Working Group (IMWG 2016) criteria. CR as negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and less than(<) 5 percent (%) plasma cells in bone marrow(BM). VGPR as serum and urine M-protein (monoclonal paraprotein) detectable by immunofixation but not on electrophoresis or 90% or greater than (>) reduction in serum and urine M-protein level <100 milligram (mg) per 24 hour (hr). PR as greater than or equal to (>=) 50% reduction of serum M-protein and less than (>=) 90% of urine M-protein or up to <200 mg per 24 hour.
Time to Next Treatment (TTNT) | Up to 3 years
  TTNT is defined as the time from the date of initiation of regimen for induction to the initiation of next regimen for each successive therapy received.
Overall Survival (OS) | Up to 3 years
  OS is defined as the time from the date of initiation of therapy to the date of death from any cause (or last documented follow-up).
Survival Time | Up to 3 years
  Survival time is defined as the time from the start of each respective treatment to death (or last documented follow-up).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score | Up to 3 years
  EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer participants. It is composed of 30 items, multiitem measure (28 items) and 2 single-item measures. For the multiple item measure, 4 point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening. The 2 single-item measure involves question about the overall health and overall quality of life which will be rated on a 7 point scale ranging from "1 = very poor" to "7 = excellent". Lower scores indicate worsening. Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Katz Index of Independence for Activities of Daily Living | Up to 3 years
  A standardized, validated tool that asks about independence in bathing, dressing, toileting, transferring, continence and feeding. The index having values from A to G. A indicates independence in all six functions and G indicates dependence in all six Functions.
Lawton Instrumental Activities of Daily Living | Up to 3 years
  This questionnaire measures participants' abilities to do instrumental activities of daily living such as ability to use telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibilities of own medication and managing finances. The scale ranges from 0 to 8, a lower scale indicates higher level of dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (69):
- United States (69):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Mercy Research, Fort Smith, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - CARTI, Little Rock, Arkansas
  - Facey Medical Group, Mission Hills, California
  - North County Oncology, Oceanside, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - James R. Berenson, MD Inc., West Hollywood, California
  - PIH Health Hospital, Whittier, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University Cancer Institute (UCI), Boynton Beach, Florida
  - Southeast Florida Hematology Oncology Group, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Watson Clinic Llp, Lakeland, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Gwinnett Hospital System, Inc, Lawrenceville, Georgia
  - Nancy N. and J.C. Lewis Cancer & Research Pavillion -St. Josephs Candler Health System, Savannah, Georgia
  - Ingalls Memorial Hospital Cancer Research Center, Harvey, Illinois
  - Orchard Healthcare Research, Skokie, Illinois
  - Baptist Healthcare Systems, Inc. d/b/a Baptist Health Floyd, New Albany, Indiana
  - Physicians' Clinic of Iowa, P.C at PCI Main Building, Cedar Rapids, Iowa
  - Commonwealth Hematology-Oncology, P.C., Danville, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Kentucky Cancer Care, Hazard, Kentucky
  - Oncology Associates of West Kentucky, Paducah, Kentucky
  - West Kentucky Hematology-Oncology, Paducah, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Tulane University Hospital & Clinics, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - MidMichigan Health Cancer Center, Midland, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - St. Luke's Speciality Clinic, Duluth, Minnesota
  - Singing River Health System, Pascagoula, Mississippi
  - Trinitas Comprehensive Cancer Center, Elizabeth, New Jersey
  - Southern Oncology Hematology Associates, Williamstown, New Jersey
  - North Shore Hematology Oncology Associates, P.C., East Setauket, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - Community Health Network, Rochester, New York
  - Mid Ohio Oncology Hematology, DBA The Mark H. Zangmeister Center, Columbus, Ohio
  - Dayton Physicians, LLC, Kettering, Ohio
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Health network (Oncology), Bethlehem, Pennsylvania
  - Hematology and Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Aria Health- Torresdale, Philadelphia, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Wellmont Blue Ridge Medical Specialists, Bristol, Tennessee
  - Jackson Madison County General Hospital, Jacksonville, Tennessee
  - Texas Oncology P A, Arlington, Texas
  - Texas Oncology P A, Beaumont, Texas
  - Texas Oncology P A, Denton, Texas
  - Texas Oncology P A, Flower Mound, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology P A, Paris, Texas
  - Texas Oncology P A, Plano, Texas
  - Texas Oncology P A, Tyler, Texas
  - Texas Oncology P A, Waco, Texas
  - Texas Oncology P A, Webster, Texas
  - Texas Oncology P A, Wichita Falls, Texas
  - Kadlec Clinic Hematology & Oncology, Kennewick, Washington